CLINICAL TRIAL: NCT06254690
Title: Safety and Efficacy of Pyrotinib in Transition From a Low-dose to Normal-dose Regimen in HER2-positive Advanced First-line Breast Cancer: a Multicenter, Open Phase II Clinical Study
Brief Title: The Dosing Regimen of Pyrotinib in HER2-positive Advanced First-line Breast Cancer: a Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Zhongda Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Jingjiang People's Hospital (Other); Yancheng First People's Hospital (Other); Affiliated Hospital of Jiangnan University (Other); Affiliated Hospital of Nantong University (Other); Anhui Provincial Cancer Hospital (Other); Huai'an First People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Suzhou Municipal Hospital (Other); Affiliated Hospital of Jiangsu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Photine
Record Dates: First submitted 2024-01-28; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: HER2 positive; Pyrotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib dose escalation group (Experimental): Pyrotinib: 240mg in the first week, 320mg in the second week, and 400mg in the third week and thereafter, by mouth(po),once a day(qd)
  Interventions: Drug: Pyrotinib dose escalation
- Pyrotinib dose normal group (Active Comparator): Pyrotinib: 400mg per week, by mouth(po),once a day(qd)
  Interventions: Drug: Pyrotinib dose normal

INTERVENTIONS:
Drug: Pyrotinib dose escalation — Pyrotinib: 240mg in the first week, 320mg in the second week, and 400mg in the third week and thereafter, by mouth(po),once a day(qd) Trastuzumab: 8mg/Kg in the first cycle, 6mg/Kg in the subsequent cycle, intravenous(iv), every 3 weeks(q3w) Docetaxel: 75mg/m2，intravenous(iv), every 3 weeks(q3w)
  Other Names: Trastuzumab; Docetaxel
  Arms: Pyrotinib dose escalation group
Drug: Pyrotinib dose normal — Pyrotinib: 400mg per week, by mouth(po),once a day(qd) Trastuzumab: 8mg/Kg in the first cycle, 6mg/Kg in the subsequent cycle, intravenous(iv), every 3 weeks(q3w) Docetaxel: 75mg/m2，intravenous(iv), every 3 weeks(q3w)
  Other Names: Trastuzumab; Docetaxel
  Arms: Pyrotinib dose normal group

SUMMARY:
Evaluate the safety and efficacy of Pyrotinib in the transition from low-dose to normal-dose regimen for HER2-positive advanced first-line breast cancer

DETAILED DESCRIPTION:
This study is planned to include 102 patients with HER2-positive advanced breast cancer meeting the admission criteria between 2023-12-01 and 2024-11-01. Statistical software will be used by the randomization officers for 1:1 allocation to pyrotinib dose increasing trial group and normal pyrotinib dose control group .

The primary endpoint of this study was grade ≥3 treatment-emergent diarrhea incidence during the first 2 cycles according to Common Terminology Criteria for Adverse Events, version 5.0, and secondary endpoints were adverse effects of pyrotinib during the study, efficacy (progression-free survival and overall survival), and patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joins the study and signs the informed consent;
2. Subject is an adult female ≥ 18 years old and ≤ 70 years old at the time of informed consent.
3. HER2-positive advanced breast cancer confirmed by pathology (HER2-positive expression refers to those with at least one tumor cell immunohistochemical staining intensity of 3+ or 2+ positive by fluorescence in situ hybridization [FISH] in the pathological examination/review of the primary or metastatic lesion conducted by the pathology department of the Central Hospital)
4. Stage IV breast cancer according to American Joint Committee on Cancer(AJCC) staging system version 8.
5. Subjects did not receive systemic antitumor therapy at the stage of recurrence/metastasis;
6. At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors version 1.1 criteria
7. When randomized, Eastern Cooperative Oncology Group(ECGO) physical fitness status is 0 or 1 point.
8. Vital organ function meets the following requirements (excluding the use of any blood components and cell growth factors during screening) : Absolute neutrophil (ANC) count ≥1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin (HB) ≥9g/dL; Serum albumin ≥3g/dL; Thyroid stimulating hormone (TSH) ≤ULN (if abnormal, T3 and T4 levels should be investigated at the same time, if T3 and T4 levels are normal, they can be included in the group); Bilirubin ≤1.5 ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN; Alkaline phosphatase (AKP) ≤ 2.5 times ULN; Serum creatinine (Cr) ≤1.5 times ULN or creatinine clearance ≥60mL/min.

Exclusion Criteria:

1. Any previous tyrosine kinase inhibitor therapy against HER2 target;
2. Patients with known active central nervous system metastases without surgery or radiation therapy, except those who have been stable for at least 1 month after treatment and have been off corticosteroids for >2 weeks;
3. Pial metastasis confirmed by MRI or lumbar puncture;
4. Inflammatory breast cancer or other malignancies within the previous 5 years, excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
5. Any antitumor therapy within 4 weeks prior to enrollment;
6. Pregnant or breastfeeding women (women of childbearing age must have a negative pregnancy test within 14 days prior to the first dose, if positive, the pregnancy must be ruled out by ultrasound);
7. Patients with gastrointestinal insufficiency or gastrointestinal disease significantly affecting the absorption of the investigational drug (e.g., uncontrolled ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or resection of the small intestine);
8. Patients with ascites, pleural effusion and pericardial effusion accompanied by clinical symptoms requiring drainage at baseline, or patients with serosal effusion drainage within 4 weeks before the first medication;
9. Patients with a history of immunodeficiency, including HIV testing positive, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
10. Patients with a major surgical procedure or significant trauma within 4 weeks before starting treatment, or expected to undergo major surgery;
11. Concomitant medical conditions (e.g., severe hypertension, diabetes, thyroid disease, co-active hepatitis B/C, and other active infections, etc.) that are deemed by the investigator to seriously endanger the patient's safety or to interfere with the patient's completion of the study;
12. Inability to understand or follow research instructions and requirements;
13. The investigator considers the patient unsuitable for entry into this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is an adult female ≥ 18 years old and ≤ 70 years old at the time of informed consent.
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of 2 cycles ≥ grade 3 diarrhea | From the date of enrollment to 2 cycles（each cycle is 28 days） of the treatment
  Grade ≥3 treatment-emergent diarrhea incidence at the end of the first 2 cycles（each cycle is 28 days） according to Common Terminology Criteria for Adverse Events(CTCAE) v5.0.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 1 year(From the date of enrollment to 30 days after the last dose)
  Adverse events include abnormal liver function, myelosuppression and so on.
Progression Free Survival | From date of randomization until the date of first documented progression from any cause, whichever came first, assessed up to 100 months
  Progression-free survival is defined as the time from the date of randomization to the date of the first documented progression as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death due to any cause.
Overall survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
Patient report outcome | through study completion, an average of 1 year(From the date of enrollment to the clinical outcome from patients' report)
  The rating is evaluated by Functional Assessment of Cancer Therapy-Breast scale. It contains questions in five dimensions, with scores ranging from 0 to 4 for each question, with higher scores generally indicating a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Yin, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No